CLINICAL TRIAL: NCT02751021
Title: Sleep Apnea Diagnosis Using a Novel Pacemaker Algorithm and Link With Aldosterone Plasma Level in Patients Presenting With Diastolic Dysfunction: SAPAAD Study
Brief Title: Sleep Apnea Diagnosis Using a Novel Pacemaker Algorithm and Link With Aldosterone Plasma Level in Patients Presenting With Diastolic Dysfunction
Acronym: SAPAAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00034-47
Record Dates: First submitted 2016-04-11; First posted 2016-04-26 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea; Arrhythmias, Cardiac; Cardiac Diastolic Function; Hyperaldosteronism
MeSH Terms: conditions — Sleep Apnea Syndromes; Arrhythmias, Cardiac; Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep apnea diagnosis (Other): The intervention is the use of the pacemaker diagnostic algorithm named Sleep Apnea Monitoring to detect sleep apnea and the attended cardiorespiratory sleep study to confirm the diagnostic.
  Interventions: Other: pacemaker diagnostic algorithm; Other: Attended cardiorespiratory sleep study

INTERVENTIONS:
Other: pacemaker diagnostic algorithm — evaluation of the respiratory disturbance index by measurement of transthoracic impedance variation, to detect sleep apnea
Other: Attended cardiorespiratory sleep study — sleep study with portable monitor resulting in the apnea hypopnea index, to confirm sleep apnea diagnosis

SUMMARY:
Little is known about potential relationships between sleep apnea, plasma aldosterone and diastolic dysfunction which is a very frequent finding among patients requiring permanent cardiac pacing. Sleep apnea is often under diagnosed by clinical examination. Confirmation tests are expensive and access is limited. A specific algorithm available in a recent pacemaker allows assessing breathing variations using minute ventilation sensor, with a good agreement between the respiratory disturbance index and polysomnography results for the diagnosis of severe sleep apnea.

The purpose of the study is to examine the diagnostic accuracy of a new pacemaker algorithm for the diagnosis of obstructive sleep apnea in patients presenting with diastolic dysfunction. The investigators also aim to highlight a correlation between plasma aldosterone levels and the severity of sleep apnea, with a reversal effect of ventilation therapy in this specific population.

ELIGIBILITY:
Inclusion Criteria:

* indication for permanent cardiac pacing (third degree atrioventricular block, second degree atrioventricular block mobitz 2 type, symptomatic sinus node dysfunction including brady-tachy form of sick sinus syndrome or bradyarrhythmia)
* Diastolic dysfunction diagnosed at the transthoracic echocardiography

Exclusion Criteria:

* younger than 18 years old
* lack of informed consent form
* impossibility to fit in the scheduled study plan
* indication for cardiac resynchronization or left ventricular ejection fraction lower than 45%
* indication for epicardial pacemaker, known severe sleep apnea treated by continuous positive airway pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Comparison between respiratory disturbance index recorded the sleep study night and Apnea hypopnea index | 2 months after pacemaker implantation
  number of apneas and hypopneas per hour (5 hours recorded by night) evaluated by the pacemaker algorithm during the night of the attended cardiorespiratory sleep study compared to the apnea hypopnea index evaluated by the portable monitor during the attended cardiorespiratory sleep study
Comparison between the mean respiratory disturbance index of the last month and Apnea hypopnea index | 2 months after pacemaker implantation
  Average value of respiratory disturbance index recorded each night during the last month compared to the apnea hypopnea index evaluated by the portable monitor during the attended cardiorespiratory sleep study

SECONDARY OUTCOMES:
Measurement of plasmatic aldosterone and correlation with apnea hypopnea index | 2 months after pacemaker implantation and one month after the beginning of continuous positive airway pressure (CPAP) therapy in apneic patients

CONTACTS AND LOCATIONS:
Overall Officials: Laure CHAMP-RIGOT, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Champ-Rigot L, Ferchaud V, Prevost JN, Moirot P, Pellissier A, Legallois D, Alexandre J, Scanu P, Morello R, Saloux E, Milliez PU. Rationale and Design for a Monocentric Prospective Study: Sleep Apnea Diagnosis Using a Novel Pacemaker Algorithm and Link With Aldosterone Plasma Level in Patients Presenting With Diastolic Dysfunction (SAPAAD Study). Clin Med Insights Cardiol. 2018 Jan 8;12:1179546817751628. doi: 10.1177/1179546817751628. eCollection 2018. PMID 29343998